CLINICAL TRIAL: NCT06826677
Title: REAL-WORLD CLINICAL OUTCOMES AMONG PATIENTS INCLUDED IN AN EARLY ACCESS PROGRAMME TREATED WITH DURVALUMAB IN COMBINATION WITH PLATINUM AND ETOPOSIDE AS FIRST-LINE THERAPY IN EXTENSIVE-STAGE SMALL CELL LUNG CANCER: AN ITALIAN MULTICENTER OBSERVATIONAL STUDY
Brief Title: REAL-WORLD DURVALUMAB IN EXTENSIVE-STAGE SMALL CELL LUNG CANCER
Acronym: ARAL
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D9070R00001
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Small Cell Lung Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — durvalumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Durvalumab — PATIENTS INCLUDED IN AN EARLY ACCESS PROGRAMME TREATED WITH DURVALUMAB IN COMBINATION WITH PLATINUM AND ETOPOSIDE AS FIRST-LINE THERAPY

SUMMARY:
Primary lung cancer is one of the most common malignancies and causes of cancer-related death worldwide [Passiglia et al., 2019; Bade and Dela Cruz, 2020].

Lung cancer is classified into different types, among which small cell lung cancer (SCLC), accounting for 13%-20% of all lung cancer cases [Pezzuto et al., 2019; Torres-Durán et al., 2021], is an aggressive form of neuroendocrine malignancy characterized by rapid growth, tendency to disseminate early and high relapse rates [El Sayed and Blais, 2021].

There are persistently limited treatment options for SCLC [DiBonaventura et al., 2019; El Sayed and Blais, 2021], and the current clinical approach to SCLC treatment is chosen irrespective of biological subtype [Rudin et al., 2021; Keogh et al., 2022]. First-line treatments for ES-SCLC have been platinum-based chemotherapy combinations for decades, without significant differences in Overall Survival (OS) between cisplatin and carboplatin, valuing flexibility in the choice of platinum agent in treatment decision making for individual patients [Dingemans et al., 2021]. However, despite the high initial response rate, the prognosis remains poor [Zhang et al., 2021; Johal et al., 2021].

In recent years, immunotherapy has dramatically modified cancer treatment across several malignancies and has been an active area of investigation in SCLC [Calles et al., 2019; Dingemans et al., 2021]. Treatments that combine chemotherapy and immune checkpoint inhibitors (ICIs), such as durvalumab and atezolizumab, can increase immune responses to tumor cells, resulting in improved efficacy in ES-SCLC compared to chemotherapy alone [Esposito et al., 2020; Konala et al., 2020; Hiddinga et al., 2021; Lim and Kang, 2021]. These treatment regimens have been approved in many countries [Wang et al., 2022] and are now the standard of care in the ES-SCLC first-line setting, according to the ESMO [Dingemans et al., 2021] and the NCCN Clinical Practice Guidelines in Oncology [Ganti et al., 2022].

Durvalumab is a fully human, immunoglobulin G1 kappa (IgG1κ) monoclonal antibody that selectively blocks the interaction of programmed cell death ligand-1 (PD-L1) with PD-1 and CD80 [IMFINZI® (durvalumab) Summary of Product Characteristics]. The phase III CASPIAN study (ClinicalTrials.gov identifier: NCT03043872) showed that the addition of durvalumab to a combination regimen of etoposide with either cisplatin or carboplatin significantly improved OS compared with etoposide and platinum alone, with a manageable tolerability profile [Paz-Ares et al., 2019; Goldman et al., 2021; Paz-Ares et al., 2022].

Following the CASPIAN study, an Early Access Programme (EAP) to provide pre-approval access to durvalumab plus platinum-etoposide for ES-SCLC patients eligible to receive first-line platinum-based chemotherapy (D419QR00007 EAP, hereafter called 'CASPIAN EAP') was activated in Italy in March 2020, including 125 subjects across 39 oncology centers.

Clinical trials have demonstrated significant efficacy and a favorable safety profile of durvalumab combined with chemotherapy in ES-SCLC [Paz-Ares et al., 2022]. On the other hand, it is estimated that stringent eligibility criteria may exclude up to 70% of patients with lung cancer from ICI clinical trials [von Itzstein et al., 2020]. Understanding the efficacy and safety of ICIs in a more heterogeneous patient population than in randomized controlled trials is critical to realizing the full potential of these therapies. To fill the gap between strictly controlled clinical trial populations and actual lung cancer patients managed in clinical practice, observational studies from real-world settings are emerging [von Itzstein et al., 2020]. Although real-world studies are unable to achieve the high internal validity of randomized controlled trials (RCTs), accurately performed analyses of real-world data can provide valuable complementary results [Nazha et al., 2021].

In conclusion, considering that ES-SCLC are often elderly patients with multiple comorbidities [Schulkes et al., 2016] for whom the treatment decision-making is challenging [DiBonaventura et al., 2019], the ARAL observational study will contribute to filling the information gap by collecting real-world data from the CASPIAN EAP to better describe durvalumab treatment outcomes and treatment patterns among patients diagnosed with ES-SCLC in Italy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with diagnosis of extensive-stage Small Cell Lung Cancer (ES-SCLC).
2. Patients entered, at least 24 months prior to the study inclusion, the D419QR00007 Early Access Programme (CASPIAN EAP) implemented in Italy.
3. Adult patients (aged ≥ 18 years) at the time of inclusion in the CASPIAN EAP.
4. Patients having performed at least one administration of durvalumab treatment in the CASPIAN EAP.
5. Patients (or their legally acceptable representatives) who have signed the subject informed consent and privacy form, if applicable.

Exclusion Criteria:

1. Patients with unavailable medical chart.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study is focused on studying a cohort of adult patients diagnosed with ES-SCLC, treated with durvalumab in combination with platinum (cisplatin or carboplatin) and etoposide as first-line therapy in the context of the CASPIAN EAP implemented in Italy. Approximately 90 subjects are expected to be included across about 15 sites in Italy, during an expected inclusion period of about 8 months.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-01-23 (Actual)

PRIMARY OUTCOMES:
Overall survival | 12 and 18 months after index date
  OS rate at 12 and 18 months after index date (defined as Day 1 of Cycle 1 - C1 D1 of platinum-etoposide chemotherapy)
Overall survival | From index date to death or date of enrollment in the study (up to 5 years)
  Median OS
Overall Survival | From index date to death or date of enrollment in the study (up to 5 years)
  Mean OS

SECONDARY OUTCOMES:
Overall Survival | 24 months after index date
  OS rate at 24 months after index date (defined as platinum-etoposide chemotherapy C1 D1).
Progression Free Survival | 12, 18, 24 months after index date
  PFS rate at 12, 18 and 24 months after index date.
Progression free survival | From index date to death or progression or date of enrollment in the study (up to 5 years)
  Median PFS
Time to discontinuation | From index date to last dose of treatment with durvalumab or death or date of enrollment in the study (up to 5 years)
  Median TTD
Time to First Subsequent Therapy or Death | From index date to start of other cancer treatment or death or date of enrollment in the study (up to 5 years)
  Median TFST
Pattern of relapse | From index date to date to progression or death or date of enrollment in the study (up to 5 years)
  Patterns of relapse after durvalumab treatment (e.g., thoracic/extra-thoracic/central nervous system - CNS relapse).
Duration of platinum-etoposide chemotherapy | From index date until durvalumab maintenance initiation or death or discontinuation of treatment (up to 5 years)
  Duration of platinum-etoposide chemotherapy prior to durvalumab maintainance initiation
durvalumab treatment duration | From initiation of durvalumab until death or date of enrollment in the study (up to 5 years)
  durvalumab treatment duration
number of durvalumab administrations | From initiation of durvalumab until death or date of enrollment in the study (up to 5 years)
  number of durvalumab administrations
reason for durvalumab dosage adjustment | From initiation of durvalumab until death or date of enrollment in the study (up to 5 years)
  reason for durvalumab dosage adjustment
reason for temporary interruption or permanent discontinuation | From initiation of durvalumab until death or date of enrollment in the study (up to 5 years)
  reason for temporary interruption or permanent discontinuation of durvalumab, (e.g., safety event)
Concomitant tratments | From initiation of durvalumab until death or date of enrollment in the study (up to 5 years)
  Details of chemotherapy (platinum-etoposide) combined with durvalumab and other concomitant treatments.
Subsequent anticancer treatments | From discontinuation of durvalumab until death or date of enrollment in the study (up to 5 years)
  Details of subsequent anticancer treatments; treatment sequences over time for ES-SCLC.
Adverse Event of Special interest (AESI)verbatim; severity; seriousness; causality; action taken with respect to durvalumab treatment; outcome. | from initiation of durvalumab until treatment discontinuation or date of enrollment in the study (up to 5 years)
  To evaluate safety and tolerability profile of durvalumab + EP treatment, adverse events of special interests were assessed. An AESI is an AE of scientific and medical interest specific to understanding of the IMP.
Adverse Event other than AESI (limited to Adverse Drug Reaction - ADR and Serious Adverse Event - SAE, including Serious Adverse Drug Reaction - SADR) verbatim; severity; seriousness; causality; action taken with respect to durvalumab treatment; outcome. | from initiation of durvalumab until treatment discontinuation or date of enrollment in the study (up to 5 years)
  To evaluate safety and tolerability profile of durvalumab + EP treatment, adverse events of special interests were assessed. An AESI is an AE of scientific and medical interest specific to understanding of the IMP.
Occurrence of at least one AESI/ ADR/ SAE/ SADR. | from initiation of durvalumab until treatment discontinuation or date of enrollment in the study (up to 5 years)
  To describe real-world safety and tolerability of durvalumab in combination with chemotherapy as first-line treatment in the CASPIAN EAP.
Durvalumab temporary interruption due to AESIs/ ADRs/SAEs/SADRs. | from initiation of durvalumab until treatment discontinuation or date of enrollment in the study (up to 5 years)
  To describe real-world safety and tolerability of durvalumab in combination with chemotherapy as first-line treatment in the CASPIAN EAP.
Durvalumab permanent discontinuation due to AESIs/ ADRs/SAEs/SADRs. | from initiation of durvalumab until treatment discontinuation or date of enrollment in the study (up to 5 years)
  To describe real-world safety and tolerability of durvalumab in combination with chemotherapy as first-line treatment in the CASPIAN EAP.

OTHER OUTCOMES:
Time interval from initial diagnosis of SCLC to test execution (e.g. biomarker test, gene mutational test,histological/cytological test) | from SCLC diagnosis to test execution (up to 3 monts)
  To describe testing patterns among patients diagnosed with ES-SCLC according to the standard clinical practice in Italy.
Time interval from diagnosis of extended disease to test execution (e.g. biomarker test, gene mutational test,histological/cytological confirmation) | from diagnosis of extended disease to test execution (up to 3 monts)
  To describe testing patterns among patients diagnosed with ES-SCLC according to the standard clinical practice in Italy.
RR | from index date until disease progression or the last evaluable assessment (up to 5 years)
  To describe the Investigator-assessed Response Rate (RR) of ES-SCLC patients treated with durvalumab plus platinum-etoposide in a real-world setting (CASPIAN EAP).

CONTACTS AND LOCATIONS:
Locations (11):
- Italy (11):
  - Research Site, Bologna
  - Research Site, Catanzaro
  - Research Site, Lucca
  - Research Site, Napoli
  - Research Site, Palermo
  - Research Site, Pistoia
  - Research Site, Prato
  - Research Site, Roma
  - Research Site, Trento
  - Research Site, Varese
  - Research Site, Vimercate

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/